CLINICAL TRIAL: NCT04965298
Title: The Effectiveness and Risks of Treating People With Idiopathic Pulmonary Fibrosis With the Addition of Lansoprazole: a Randomised Placebo-controlled Multi-centre Clinical Trial
Brief Title: Treating People With Idiopathic Pulmonary Fibrosis With the Addition of Lansoprazole
Acronym: TIPAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: Norwich Clinical Trials Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 269050-80-06-19; 2020-000041-14 (EudraCT Number); 269050 (Other: IRAS number); ISRCTN13526307 (Other: ISRCTN number)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; IPF; Lansoprazole; Proton pump inhibitors; Cough; FVC; Forced vital capacity; Domiciliary spirometry; Virtual clinical trial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Lansoprazole

STUDY DESIGN:
Intervention Model Description: This study is an interventional clinical trial of an investigational medicinal product: a phase III, randomised, placebo-controlled, two arm parallel group, double-blind, multicentre clinical trial.
  Randomisation will be generated by a secure web-based system on a 1:1 basis with minimisation for recruiting site, baseline IPF treatment, reflux and cough.
  All study visits may be conducted remotely without the need for participants to attend the participating site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator, outcomes assessor. Statistician. Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment arm (Experimental): Lansoprazole 30mg (as 2 x 15mg capsules) twice daily, 12 hours apart, for 12 months. IMP should be taken at least 30 minutes before food.
  Interventions: Drug: Lansoprazole
- Matched-Placebo arm (Placebo Comparator): Matched placebo 2 capsules twice daily, 12 hours apart, for 12 months. Treatment should be taken at least 30 minutes before food.
  Interventions: Other: Matched placebo

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30mg (as 2 x 15mg capsules) twice daily, 12 hours apart, for 12 months. IMP should be taken at least 30 minutes before food.
  Arms: Active treatment arm
Other: Matched placebo — Matched placebo 2 capsules twice daily, 12 hours apart, for 12 months. Treatment should be taken at least 30 minutes before food.
  Arms: Matched-Placebo arm

SUMMARY:
IPF is a progressive scarring lung condition causing coughing and breathlessness. IPF patients often have reflux disease meaning stomach acid may be breathed into the lungs, potentially damaging them. Medicines which stop stomach acid production, proton pump inhibitors (PPIs), can be used to reduce reflux symptoms including heartburn. Some researchers suggest PPIs also reduce IPF progression.

This research aims to see if IPF progresses slower if treated with PPIs. Based on the results, we will be able to recommend whether or not IPF patients should take PPIs.

This trial will involve 298 IPF patients from approximately 37 UK hospitals. At the beginning of the study, we will ask patients to start performing weekly breathing tests at home using equipment provided, and ask those with a cough to use a device to count the number of times they cough in 24hours. We will ask them to answer two questions rating their coughing and breathlessness, and complete questionnaires on their coughing, IPF, sleep habits and general condition. People will be given a PPI, called lansoprazole, or dummy tablets, twice per day for 12 months. They will be given a leaflet telling them what to do about reflux symptoms. At the end of the study, we will repeat these tests and analyse the results. We will record any side effects people may get. If people suffer side effects, they can reduce the dose.

People taking medicines that interact with PPIs or have other serious medical conditions won't be able to participate. People receiving PPIs will only be able to participate if they can stop taking their medication without their heartburn returning.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive and usually fatal lung disease with a poor prognosis. IPF patients frequently have other medical conditions as well, with reflux disease being one of the most common. Previous studies and a review of data already collected suggest that treatments used to reduce reflux disease symptoms, proton pump inhibitors (PPIs), may reduce IPF disease progression and improve survival rates. Current IPF treatment guidelines cautiously advise PPI treatment for IPF patients, however there hasn't been a study which investigates this specifically yet even though doctors and government groups have said one is needed. There are thought to be links between cough, reflux, sleep and IPF. As a result we will be asking a sub-group of patients to complete two 24 hour sessions of cough frequency monitoring as a sub-study. Some of these participants may be asked to wear a wrist-based activity and sleep monitor during these periods also. In addition, we will ask patients to complete two questionnaires on their sleeping habits to further investigate this link. At the end of the trial, we will able to recommend whether or not IPF patients should take PPIs routinely or not.

This project is a clinical trial of an investigational medicinal product (drug). The drug is well established and approved for use for another medical condition. The drug will be assessed against placebo (dummy) tablets, with patients allocated to either group by chance. Patients on the drug and dummy tablets will be assessed at the same time. Neither patients nor their doctors or the research team will know which treatment they have been allocated to. We will be running the study at approximately 37 hospitals across the UK.

All study visits may take place remotely without the participant needing to attend the hospital. However, face-to-face onsite visits are also permitted if preferred/feasible. All participants will receive central training via video call, with a trained clinical physiologist, following consent on how to complete domiciliary spirometry assessments. Further training will be provided during follow-up if deemed required following a review of the data. Questionnaires will be completed either electronically or by post.

Potentially eligible patients will be approached remotely or in clinic after being identified from local patient lists/databases. They will be given/sent the relevant study literature to consider participation in the study and will be followed-up by a member of the local research team after they have had at least 24hours to consider participating.

Interested patients will be invited to a virtual or face-to-face screening appointment where they will be counselled on the study and what it entails in order to provide informed consent to participate. The patient will then be asked to complete baseline questionnaires, provide demographic, medical history and concomitant medication, and any other relevant study information, complete spirometry assessments over 5 days at home using a domiciliary spirometer and provide a blood sample for safety in order for the investigator to confirm their eligibility for the trial. Patients may also provide a blood sample for analysis in future research if the visit takes place at the recruiting site. In addition, eligible participants may complete a 24hour period of cough frequency monitoring, and activity and sleep monitoring if applicable, if they have consented to do so. Patients in receipt of PPIs without a clear clinical indication for them at consent, will undergo a two week wash-out period (following agreement from the patient and their GP) to ascertain whether it is safe to stop this treatment and monitor whether their symptoms subside. Patients who remain asymptomatic at the end of this period will proceed to enter the study. For those whose symptoms return, PPI treatment will recommence and they will not enter the study. Once the results of all baseline assessments are known, patients will be randomised.

Participants will receive an initial 6 month supply of trial medication and be instructed to take 2 tablets twice daily (approximately 12 hours apart), 30 minutes before meals, for 12 months. Participants will commence weekly domiciliary spirometry assessments, for 12 months, from this point onwards.

At 3 months post-randomisation, participants will complete the relevant questionnaires and provide blood samples for safety checks. Domiciliary spirometry assessments remain ongoing. Participants involved in the sub-study will again undergo cough frequency monitoring, and activity and sleep monitoring if applicable, for a final 24 hour period. Patients will be asked to report any changes in their medical history, medication and any events which they have experienced since their last visit.

Participants will be contacted again at 6 months post-randomisation where they we will complete questionnaires and provide a safety blood samples. Domiciliary spirometry assessments remain ongoing. Participants will again be asked to report any changes in their medical history, medication and any events which they have experienced since their last visit. Participant adherence to the trial medication will be checked. A final supply of trial medication will be dispensed.

At 9 months post-randomisation, local site staff will contact patients to record any changes in their medical history, medication and any events experienced since their last visit. Patients will be required to complete the required questionnaires and provide a blood sample for safety checks.

The final study assessments will be at 12 months post-randomisation. Patients will be required to complete all necessary questionnaires, provide a blood sample for safety analysis and a final set of domiciliary spirometry assessments will occur over a 5 day consecutive period. If participants have consented to do so, an additional blood sample will be taken for analysis in future research studies if the visit occurs on site. Patients will be required to report any changes in their medical history, medication and any events they have experienced since their last report to site staff.

If participants are suspected of or confirmed to have experienced any of the following they may reduce the dose of their trial treatment, at any point during the study, to 1 tablet, twice daily (approximately 12 hours apart), 30 minutes before meals: infection including pneumonia, Clostridium difficile infection and/or hypomagnesaemia. Participants may also reduce dose if the participant or clinician wishes them to do so.

A blood sample for genotype analysis may be taken at any study timepoint which occurs face-to-face, if the participants consents to provide one. Safety blood samples will be taken at the participant's GP surgery where visits take place remotely. Remote follow-up may take place via video or phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged greater than or equal to 40 years.
2. A diagnosis of Idiopathic Pulmonary Fibrosis (IPF) based on local or regional multi-disciplinary consensus according to the latest international guidelines (50).
3. Patients may be receiving licensed anti-fibrotic medication (for at least 4 weeks prior to randomisation with no planned amendments for at least 4 weeks post-randomisation).
4. Able to provide informed consent.

Additional Inclusion Criteria for cough count sub-study:

1. Pre-existing diagnosis of persistent cough (defined as troublesome for more than 8 weeks prior to study enrolment).

Exclusion Criteria:

1. Patients unable to comply with study assessments including the ability to complete reliable spirometry assessments.
2. Concomitant use of a proton pump inhibitor (PPI) or prokinetic drugs (cisapride, domperidone, metoclopramide, erythromycin, prucalopride etc.) within 2 weeks prior to randomisation.
3. Patients with a self-reported respiratory tract infection within 4 weeks of screening (defined as two or more of: increased cough, sputum or breathlessness and requiring antimicrobial therapy).
4. Significant co-existing respiratory disease (defined as a respiratory condition that exhibits a clinically relevant effect on respiratory symptoms and disease progression as determined by the PI). The presence of traction bronchiectasis is permitted.
5. Patients with an FEV1/FVC<0.7.
6. Significant medical, surgical or psychiatric disease that in the opinion of the patient's attending physician would affect subject safety or influence the study outcomes including liver failure (e.g. serum transaminase > 2 x upper limit of normal (ULN), Bilirubin > 1.5 x ULN (unless the patient has Gilbert's Syndrome) and chronic kidney disease (CKD) greater than stage 3 , erosive oesophagitis, Barrett's oesophagus or any condition requiring lifelong proton pump inhibitor use.
7. Known allergy to proton pump inhibitors or the contents of placebo.
8. Concomitant use of atazanavir, ketoconazole, itraconazole, tacrolimus, methotrexate, fluvoxamine (see section 6.4.5).
9. Females who are of childbearing potential or lactating. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
10. Receipt of another investigational drug or biological agent associated with another clinical trial within the 4 weeks prior to TIPAL study enrolment or 5 times the drug half-life, whichever is the longer.
11. Receiving long-term oxygen therapy.
12. Patients with hypomagnesemia (defined as magnesium ≤0.6 mmol/L).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Absolute change in percent predicted (%) forced vital capacity (FVC) | 12 months post-randomisation
  Absolute change in percent predicted (%) forced vital capacity (FVC) at 12 months post-randomisation of lansoprazole versus placebo.

SECONDARY OUTCOMES:
Cough frequency | 3 months post-randomisation
  Cough frequency measured using a VitaloJAK cough monitor over a 24h period.
Cough score | 3, 6, 9 and 12 months post-randomisation
  Cough score measured using a 100mm visual analogue scale (VAS).
Cough related | 3, 6, 9 and 12 months post-randomisation
  Cough related quality of life measured by the Leicester Cough Questionnaire (LCQ).
Breathlessness | 3, 6, 9 and 12 months post-randomisation
  Breathlessness measured by the Medical Research Council Dyspnoea scale.
Disease specific quality of life | 3, 6, 9 and 12 months post-randomisation
  Disease specific quality of life measured using the King's Brief Interstitial Lung Disease (K-BILD) questionnaire.
Health related quality of life | 3, 6, 9 and 12 months post-randomisation
  Health related quality of life measured using the EQ-5D-5L questionnaire (quality adjusted life years will be estimated).
Total lung diffusing capacity of carbon monoxide | 3, 6 and 12 months post-randomisation
  Total lung diffusing capacity of carbon monoxide (DLCO) measured (corrected for haemoglobin) where possible.
Laboratory assessment | 3, 6 and 12 months post-randomisation
  Laboratory assessment of FVC and FEV1 where possible.
Sleep quality | 3 and 12 months post-randomisation
  Sleep quality measured by the short Pittsburgh Sleep Quality Index (PSQI).
Reflux characteristics | 3 and 12 months post-randomisation
  Reflux characteristics measured by the DeMeester score.
Participant acceptability | 12 months post-randomisation
  Participant acceptability measured by a study-specific questionnaire.
Risk of sleep apnoea | 12 months post-randomisation
  Risk of sleep apnoea measured by the STOP-Bang questionnaire.
Progression free survival | 12 months post-randomisation
  Progression free survival (with progression defined as time from date of randomisation to week of all-cause death, lung transplant or a 10% absolute reduction in FVC % predicted from baseline measured by weekly domiciliary spirometry).
Hospital-free survival defined as death | 12 months post-randomisation
  Hospital-free survival defined as death (all-cause) or first non-elective (all-cause) hospital admission.
Respiratory related hospital free survival | 12 months post-randomisation
  Respiratory related hospital free survival.
The decline and rate of decline in absolute %FVC | Measured over the course of 12 months
  The decline and rate of decline in absolute %FVC based on %FVC measured weekly by domiciliary spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Andrew Wilson, Study Chair — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (57):
- United Kingdom (57):
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - NHS Grampian, Aberdeen
  - Northern Health and Social Care Trust, Antrim
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - University Hospitals Birmingham NHS Foundation Trust (QEHB), Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - East Lancashire Hospitals NHS Trust, Blackburn
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - North Bristol NHS Trust, Bristol
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - Hywel Dda University Health Board, Carmarthen
  - Southern Health & Social Care Trust, Craigavon
  - Mid Cheshire Hospitals NHS Foundation Trust, Crewe
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - NHS Tayside, Dundee
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Frimley Health NHS Foundation Trust, Frimley
  - The Princess Alexandra Hospital NHS Trust, Harlow
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - Hull University Teaching Hospitals NHS Trust, Hull
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Kendal
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Western Health and Social Care Trust, Londonderry
  - Bedfordshire Hospitals NHS Foundation Trust, Luton
  - East Cheshire NHS Trust, Macclesfield
  - Manchester University NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - East and North Hertfordshire NHS Trust, Stevenage
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - University Hospitals of North Midlands, Stoke-on-Trent
  - South Tyneside And Sunderland NHS Foundation Trust, Sunderland
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Somerset NHS Foundation Trust, Taunton
  - Kingston and Richmond NHS Foundation Trust, Teddington
  - Torbay and South Devon NHS Foundation Trust, Torquay
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan
  - The Royal Wolverhampton NHS Trust, Wolverhampton
  - Worcestershire Acute Hospitals NHS Trust, Worcester
  - York and Scarborough Teaching Hospitals NHS Foundation Trust, York

REFERENCES:
- [Derived] Jones M, Cahn A, Chaudhuri N, Clark AB, Forrest I, Hammond M, Jones S, Maher TM, Parfrey H, Raghu G, Simpson AJ, Smith JA, Spencer LG, Thickett D, Vale L, Wahed S, Ward C, Wilson AM. The effectiveness and risks of Treating people with Idiopathic Pulmonary fibrosis with the Addition of Lansoprazole (TIPAL): study protocol for a randomised placebo-controlled multicentre clinical trial. BMJ Open. 2025 Feb 5;15(2):e088604. doi: 10.1136/bmjopen-2024-088604. PMID 39909521

DOCUMENTS (1):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04965298/Prot_001.pdf